CLINICAL TRIAL: NCT01683708
Title: Effectiveness of Perioperative Symbiotic Therapy to Reduce Infectious Morbidity in Jaundiced Patients: a Randomized Controlled Trial
Brief Title: Effectiveness Of Symbiotic Therapy In Jaundiced Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Ordine Mauriziano di Torino (Other)
Responsible Party: Principal Investigator, LorenzoCapussotti, Director of Department of General and Oncologica Surgery, Azienda Ospedaliera Ordine Mauriziano di Torino
Other Study IDs: Symbiotic2012
Record Dates: First submitted 2012-09-07; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Postoperative Infections; Jaundice
Keywords: sepsis; jaundice; symbiotic; translocation; abdominal collection; morbidity
MeSH Terms: conditions — Jaundice; Sepsis | interventions — Prebiotics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Symbiotic group: Jaundiced patients who have symbiotic therapy
  Interventions: Dietary Supplement: Symbiotic therapy
- No Symbiotic therapy: Jaundiced patients who not have symbiotic therapy

INTERVENTIONS:
Dietary Supplement: Symbiotic therapy — Patients randomized into the Symbiotic group received Prebiotic® in a dose of one sachet twice a day for at least 1 week preoperatively. Postoperatively the medication was reintroduced as tolerated, and continued until discharge from hospital. One 4,5 gr sachet of Prebiotic® contains at least 1010 living Bifidobacterium bifidum, 1010 living Streptococcus Thermophilus, 1010 living Streptococcus Salivarius, 3 109 Lactobacillus Acidophilus, 1010 living Lactobacillus Casei, 1010 living Lactobacillus bulgaricus and galactooligosaccharides (4,5 gr).
  Other Names: Prebiotic® (Mediabase s.r.l., Prato, Italy)
  Groups: Symbiotic group

SUMMARY:
The aim of the present study was therefore to evaluate if the perioperative administration of symbiotics reduces postoperative infectious morbidity in jaundiced patients scheduled for hepato-biliary and pancreatic surgery.

DETAILED DESCRIPTION:
Despite advances in preoperative patient's selection and anesthetic and surgical techniques, surgery in jaundiced patients is associated with significant morbidity and mortality as a consequence of septic complications. The evidence that nosocomial infections are frequently a consequence of gut-derived organism such as enterobacteriaceae, supports the hypothesis of the "gut derived sepsis". Indeed, several studies have reported that jaundiced patients present an increased intestinal permeability and consequently a higher rate of bacterial migration from gastrointestinal tract across the lamina propria to local mesenteric lymph nodes and from there to extra-intestinal site. This phenomenon increases after surgical decompression of bile duct. The higher prevalence of bacterial translocation in jaundiced patients is related to different mechanisms such as mucosal atrophy secondary to protracted absence of intraluminal bile that open para-cellular route for bacterial translocation and the decreased clearance capacity of Kuppfer secondary to cholestasis.

The mechanisms of action of symbiotics are largely unknown. The probiotic bacteria can improve the mucosal barrier function reducing the bacterial translocation of organism to mesenteric lymph nodes. Indeed symbiotic can affect the intestinal ecosystem by stimulating mucosal immune and non-immune mechanisms through antagonism/competition with potential pathogens.

ELIGIBILITY:
Inclusion Criteria:

* jaundiced patients scheduled for elective extrahepatic bile duct resections
* age between 18 and 80 year-old Exclusion Criteria:

Exclusion Criteria

* cirrhosis
* American Society of Anesthesiologists (ASA) score 4
* intestinal malabsorption
* emergency surgery
* intolerance to symbiotic
* diagnosis of primary or secondary immunodeficiency
* unresectability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Jaundiced patients scheduled for hepato-biliary pancreatic surgery
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-11

PRIMARY OUTCOMES:
Infectious Morbidity Rate | Participants will followed for the duration of hospital stay, an expected average of 6 weeks

SECONDARY OUTCOMES:
IMMUNE PROFILE | The day before and on postoperative day 7
RATE OF TRANSLOCATION | Intraoperative
  a lymph node was routinely excised from the ileocaecal mesentery and was immediately transported in sterile saline to the laboratory for culture

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Capussotti, MD, Principal Investigator — Mauriziano Hospital, Department of General and Oncological surgery

REFERENCES:
- [Result] Sugawara G, Nagino M, Nishio H, Ebata T, Takagi K, Asahara T, Nomoto K, Nimura Y. Perioperative synbiotic treatment to prevent postoperative infectious complications in biliary cancer surgery: a randomized controlled trial. Ann Surg. 2006 Nov;244(5):706-14. doi: 10.1097/01.sla.0000219039.20924.88. PMID 17060763
- [Result] Kanazawa H, Nagino M, Kamiya S, Komatsu S, Mayumi T, Takagi K, Asahara T, Nomoto K, Tanaka R, Nimura Y. Synbiotics reduce postoperative infectious complications: a randomized controlled trial in biliary cancer patients undergoing hepatectomy. Langenbecks Arch Surg. 2005 Apr;390(2):104-13. doi: 10.1007/s00423-004-0536-1. Epub 2005 Feb 12. PMID 15711820